CLINICAL TRIAL: NCT04275544
Title: Perioperative Risk Factors of Postoperative Complications in Hypertrophic Obstructive Cardiomyopathy Patients Undergoing Septal Myectomy
Brief Title: Risk Factors of Postoperative Complications in HCM Patients
Acronym: RFHCM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, chonglei, Clinical professor, Xijing Hospital
Other Study IDs: KY20200121-C-1
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Hypertrophic Obstructive Cardiomyopathy; Risk factor; Postoperative complication
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with PCs: HOCM Patients developing postoperative complications (PCs) following septal myectomy.
  PCs include all-cause mortality, heart failure, low cardiac output syndrome, stroke, spinal cord injury, acute respiratory distress syndrome, reintubation, reoperation, permanent implantable cardioverter defibrillator, kidney injury, renal failure, liver injury, and liver failure.
- Patients without PCs: HOCM Patients do not develope postoperative complications following septal myectomy.

SUMMARY:
Perioperative management may have strong connections with postoperative complications (PCs). However, little is known about the perioperative risk factors of PCs after septal myectomy in hypertrophic obstructive cardiomyopathy (HOCM) patients. This study is designed to assess the in-hospital PCs rate of HOCM patients and to identify perioperative risk factors of PCs in patients who underwent septal myectomy. Retrospective chart review will identify adult HOCM patients who underwent septal myectomy from October 2013 to December 2018 in the investigators' hospital. Patients' data will be collected from electronic medical records. The multivariable logistic regression analysis will be used to determine independent predictors. The predictive ability of individual predictor and different combination of multiple risk factors on PCs will also be calculated.

DETAILED DESCRIPTION:
This study is a single center retrospective observational study designed to assess the in-hospital PCs rate of HOCM patients and to identify perioperative risk factors of PCs in patients who underwent septal myectomy.

Ethical approval of this study was obtained from the Institutional Review Board of the investigators' hospital (No. KY20192036-C-1). The requirement for written informed consent was waived by the Institutional Review Board, considering the retrospective nature of the study.

Retrospective chart review will identify adult HOCM patients who underwent septal myectomy from October 2013 to December 2018 in the investigators' hospital. The clinical diagnosis of HOCM is made by echocardiography, cardiac magnetic resonance imaging, or computed tomography of a hypertrophied, non-dilated LV, in the absence of cardiac or systemic disease that can aggravate the magnitude of hypertrophy.

Data Collection

The following data will be collected. Data will be obtained from electronic medical records and collected by two trained staff who are unaware of the purpose of the study.

1. Demographic and clinical data included New York Heart Association class, family history of hypertrophic cardiomyopathy (HCM) and sudden death, patient history, symptoms, medications, and comorbidities of these enrolled patients.
2. The following preoperative echocardiographic parameters will be collected : left atrium diameter, left ventricular (LV) ejection fraction (EF), maximal LV wall thickness (defined as the greatest thickness measured at any site within the LV wall), maximal interventricular septal thickness, left ventricular outflow tract diameter (LVOTd) (C-sept distance, the shortest distance from the septum to the coaptation point of the mitral valve), and resting left ventricular outflow tract (LVOT) gradient (measured with continuous-wave Doppler in the apical five-chamber view using the modified Bernoulli equation).
3. Intraoperative data collected include the duration of anaesthesia, surgery, CPB, and cross-clamp; excised LV weight; type of concomitant procedure; lowest body temperature, haematocrit , haemoglobin and highest Lactic acid; perioperative fluid management including the volumes of total fluid intake, total output and intraoperative fluid balance (total intraoperative fluid intake is calculated as the sum of crystalloid, colloid and blood products; total output was calculated as the sum of the volumes of estimated blood loss and urine output; intraoperative fluid balance is calculated by subtracting the total output from the total fluid intake); and blood pressure parameters including the baseline mean arterial pressure and lowest mean arterial pressure, and duration of intraoperative hypotension (intraoperative hypotension is defined as a mean arterial pressure <65 mmHg).
4. Postoperative ventilation hours, lengths of stay in the intensive care unit (ICU) and hospital, blood transfusion in 72 hours after surgery, EF, LVOTd, resting LVOT gradient gradient, and in-hospital PCs will also be obtained. In-hospital PCs include all-cause mortality, heart failure, low cardiac output syndrome, stroke, spinal cord injury, acute respiratory distress syndrome, reintubation, reoperation, permanent implantable cardioverter defibrillator, kidney injury, renal failure, liver injury, and liver failure.

Statistical analysis

Continuous variables will be expressed as mean ± standard deviation (SD) or median (interquartile range). Differences of continuous variables will be analysed by using a parametric unpaired Student's t-test or non-parametric Mann-Whitney U-test, as appropriate. Categorical variables will be described as percentages (%) and compared using the chi-square test or Fisher's exact test. For all analyses, a two-tailed P-value <0.05 will be considered statistically significant. The multivariable model will be used to determine independent predictors by including only variables that are identified by univariable analysis as significant prognosis risk factors with a P-value <0.05. Receiver operating characteristic curve will be used to calculate the cut off values of individual risk factors. The predictive ability of individual predictor and different combination of multiple risk factors on PCs will also be calculated. SPSS software version 22.0 (IBM Corp., Armonk, NY, USA) will be used to analyse the data.

Privacy

All data collected in this study will be stored on computer systems that require user authentication for log on. After data collection is complete, none of this electronic data will be stored with subject-identifying information and will be archived and kept indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of age who underwent thoracotomy for septal myectomy.

Exclusion Criteria:

* Patients with severe liver and renal disease, severe central nervous system disease, malignancy, defibrillators and age under 18 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed clinical diagnosis of HOCM were referred for surgical septal myectomy in a tertiary hospital in China
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Identify perioperative risk factors of in-hospital postoperative complications (PCs) | From the surgery start to patient discharge from hospital, normally within 20 days
  Identify the perioperative risk factors of in-hospital PCs by multivariable logistic regression analysis.
  Intraoperative data collected include the duration of anaesthesia, surgery, CPB, and cross-clamp; excised LV weight; type of concomitant procedure; lowest body temperature, haematocrit , haemoglobin and highest Lactic acid; perioperative fluid management including the volumes of total fluid intake, total output, blood loss and urine output; and blood pressure parameters including the baseline mean arterial pressure and lowest mean arterial pressure, and duration of intraoperative hypotension (intraoperative hypotension was defined as a mean arterial pressure <65 mmHg).
  In-hospital PCs include all cause mortality, heart failure, low cardiac output syndrome, stroke, spinal cord injury, acute respiratory distress syndrome, reintubation, reoperation, permanent implantable cardioverter defibrillator, kidney injury, renal failure, liver injury, and liver failure.

SECONDARY OUTCOMES:
The incidence of in-hospital postoperative complications (PCs) | From the end of surgery to patient discharged from hospital, normally within 20 days
  In-hospital PCs include all cause mortality, heart failure, low cardiac output syndrome, stroke, spinal cord injury, acute respiratory distress syndrome, reintubation, reoperation, permanent implantable cardioverter defibrillator, kidney injury, renal failure, liver injury, and liver failure.

OTHER OUTCOMES:
Hospital-stay | During patient stay in hospital, normally within 30 days
  The number of days patient stay in hospital
ICU-stay | From the end of surgery to patient discharged from ICU, normally within 10 days
  The number of days patient stay in ICU after surgery
Postoperative mechanical ventilation | From the end of surgery to tracheal extubation, normally within 48 hours
  Duation of postoperative mechanical ventilation
Postoperative hospital stay | From the end of surgery to patient discharged from hospital, normally within 20 days
  Length of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, MD, Ph.D, Study Director — Director of the Department of Anesthesiology and Perioperative Medicine
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Background] Brown ML, Schaff HV. Surgical management of obstructive hypertrophic cardiomyopathy: the gold standard. Expert Rev Cardiovasc Ther. 2008 Jun;6(5):715-22. doi: 10.1586/14779072.6.5.715. PMID 18510487
- [Background] Parry DJ, Raskin RE, Poynter JA, Ribero IB, Bajona P, Rakowski H, Woo A, Ralph-Edwards A. Short and medium term outcomes of surgery for patients with hypertrophic obstructive cardiomyopathy. Ann Thorac Surg. 2015 Apr;99(4):1213-9. doi: 10.1016/j.athoracsur.2014.11.020. Epub 2015 Feb 10. PMID 25678500
- [Background] Desai MY, Bhonsale A, Smedira NG, Naji P, Thamilarasan M, Lytle BW, Lever HM. Predictors of long-term outcomes in symptomatic hypertrophic obstructive cardiomyopathy patients undergoing surgical relief of left ventricular outflow tract obstruction. Circulation. 2013 Jul 16;128(3):209-16. doi: 10.1161/CIRCULATIONAHA.112.000849. Epub 2013 Jun 14. PMID 23770748
- [Background] Woo A, Williams WG, Choi R, Wigle ED, Rozenblyum E, Fedwick K, Siu S, Ralph-Edwards A, Rakowski H. Clinical and echocardiographic determinants of long-term survival after surgical myectomy in obstructive hypertrophic cardiomyopathy. Circulation. 2005 Apr 26;111(16):2033-41. doi: 10.1161/01.CIR.0000162460.36735.71. Epub 2005 Apr 11. PMID 15824202
- [Background] Tang B, Song Y, Cui H, Ji K, Zhu C, Zhao S, Huang X, Yu Q, Hu S, Wang S. Prediction of Mid-Term Outcomes in Adult Obstructive Hypertrophic Cardiomyopathy After Surgical Ventricular Septum Myectomy. J Am Coll Cardiol. 2017 Oct 17;70(16):2092-2094. doi: 10.1016/j.jacc.2017.08.032. No abstract available. PMID 29025563
- [Derived] Fan Q, Lu Z, Wang Y, Wang L, Zhang H, Zheng Z, Dong H, Xiong L, Lei C. Association between postoperative nadir platelet count and postoperative cardiovascular complications following septal myectomy in patients with hypertrophic cardiomyopathy: a retrospective cohort study. BMC Cardiovasc Disord. 2024 Jan 18;24(1):57. doi: 10.1186/s12872-024-03724-2. PMID 38238666